CLINICAL TRIAL: NCT07385105
Title: Exploring Cognitive Behavioral Therapy for Insomnia (CBT-I) in Mild Traumatic Brain Injury (mTBI)
Brief Title: Evaluation of Cognitive Behavioral Therapy for Insomnia (CBT-I) in Individuals With Mild Traumatic Brain Injury (mTBI)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Sepideh Zenoozi, PhD candidate, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2131848
Record Dates: First submitted 2026-01-11; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Sleep Architecture; Mild Traumatic Brain Injury; Sleep; Sleep and Circadian Problems
Keywords: Sleep problems; Cognitive behavioral Therapy for insomnia; CBT-I; mild traumatic brain injury; mTBI; Functional performance
MeSH Terms: conditions — Brain Concussion; Parasomnias | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: All participants will receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 15 mTBI cases who have sleep problems will receive CBT-I (Experimental): We will achieve the study's aims with a single-group, pre-post design (n=15). Participants with physician-diagnosed mild traumatic brain injury who are experiencing sleep problems for more than four weeks will receive cognitive behavioral therapy for insomnia (CBT-I). Participants will engage in six one-hour, weekly CBT-I sessions delivered in a one-on-one format through the Zoom Video Conference. Participants will establish sleep-related goals. During the intervention session, the interventionist will address the cognitive and behavioral components of CBT-I, as well as relaxation techniques and sleep hygiene.
  Interventions: Behavioral: Cognitive behavioral Therapy for insomnia (CBT-I)

INTERVENTIONS:
Behavioral: Cognitive behavioral Therapy for insomnia (CBT-I) — CBT-I is an evidence-based psychotherapy designed to address insomnia. This structured and multifaceted intervention aims to help individuals who have trouble falling asleep or/ and staying asleep during the night. CBT-I is a multi-component treatment that includes two core parts: behavioral and cognitive aspects. It consists of Sleep Restriction Therapy (SRT), Stimulus Control Therapy (SCT), and Cognitive Therapy (CT) with an emphasis on Cognitive restructuring, as well as Psychoeducation and Sleep Hygiene Education. Each CBT-I session has a clear structure and includes various components such as assessment, psychoeducation, behavioral and cognitive interventions, adherence monitoring, and strategies for preventing relapse. In this study, participants will receive CBT-I in a one-on-one setting, meeting on Zoom once a week for six weeks, and each session will last an hour.

SUMMARY:
This study will employ cognitive behavioral therapy for insomnia (CBT-I) among individuals with mild traumatic brain injury (mTBI) who experience sleep disturbances. The research aims to evaluate the effects of CBT-I on sleep, mTBI symptoms, and, in particular, the ability of individuals with mTBI to engage in their desired daily life activities. The main questions this study aims to answer are:

1. Does CBT-I positively impact symptoms of mTBI?
2. Does CBT-I improve functional performance in individuals with mTBI?

DETAILED DESCRIPTION:
Cognitive behavioral therapy for insomnia (CBT-I) is an evidence-based intervention that has demonstrated significant results in various populations. CBT-I is a structured and goal-oriented approach that addresses both unhelpful thoughts and maladaptive behaviors contributing to poor sleep. CBT-I includes several components, such as behavioral strategies that aim to change habits disrupting sleep architecture and cognitive techniques targeting maladaptive beliefs about sleep. However, limited research has examined the use of this intervention among individuals with mild traumatic brain injury (mTBI), particularly regarding its impact on their ability to perform daily life activities. This study aims to evaluate how CBT-I can impact sleep, mTBI symptoms, and participants' functional performance.

ELIGIBILITY:
Inclusion Criteria:

* A history of mTBI documented by a physician and sleep problems for more than 4 weeks
* A score ≥ 10 on the Insomnia Severity Index (ISI)
* Speak, read, and write English

Exclusion Criteria:

* History of other neurological or psychological conditions
* Patient Health Questionnaire-9 (PHQ-9) score higher than 20 (severe depressive symptoms)
* Generalized Anxiety Disorder-7 (GAD-7) score higher than 15 (severe anxiety symptoms)
* Montreal Cognitive Assessment (MoCA) score less than 24

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The expanded consensus sleep diary (CSD) | Through study completion, an average of 10 weeks.
  The expanded consensus sleep diary (CSD) is intended for use both in the morning and evening. Participants are required to complete the diary each morning upon waking and each evening before bedtime. The evening section records information about daytime activities, including caffeine, alcohol, medication use, and napping. The morning section captures details regarding the previous night's sleep.
Insomnia Severity Index (ISI) | Baseline (Day 1)
  The Insomnia Severity Index (ISI) is a seven-item questionnaire developed to assess the severity of insomnia symptoms. Scores range from 0 to 28, with higher scores indicating more severe symptoms.
Pittsburgh Sleep Quality Index (PSQI) | Baseline (Day 1)
  The Pittsburgh Sleep Quality Index (PSQI) is a sleep questionnaire that evaluates seven primary components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction over a one-month period. The PSQI is used to assess the impact of cognitive behavioral therapy for insomnia (CBT-I) on these sleep components. Scores range from 0 to 21, with higher scores indicating poorer sleep quality.
Epworth Sleepiness Scale (ESS) | Baseline (Day 1)
  The Epworth Sleepiness Scale (ESS) is a sleep questionnaire consisting of 8 items that assesses daytime sleepiness. A score of 10 or higher indicates pathological daytime sleepiness. The total score ranges from 0 to 24, with higher scores indicating greater daytime sleepiness.
Canadian Occupation Performance Measure (COPM) | Baseline (day 1)
  The Canadian Occupation Performance Measure (COPM) is a self-reported measure of an individual's perceived performance and satisfaction in important daily activities. Scores range from 1 (low) to 10 (high) for both performance and satisfaction, with higher scores indicating better outcomes.
Activity Card Sort (ACS) | Baseline (day 1)
  Occupational therapists use the Activity Card Sort (ACS) to help clients describe their social, instrumental, and leisure activities. For this study, we are going to use Electronic Activity Card Sort. It serves the same purpose as the paper/card version but is administered electronically. Total scores are expressed as a percentage (0-100%), with higher scores indicating greater participation and activity engagement.
Feasibility of Intervention Measure (FIM) | Post intervention (final study visit)
  Feasibility of Intervention Measure (FIM) is a questionnaire that includes 12 items for evaluating acceptability, feasibility, and appropriateness of the Intervention.
Client Satisfaction Questionnaire (CSQ-8) | Post intervention (final study visit)
  The Client Satisfaction Questionnaire (CSQ-8) was used to evaluate participant satisfaction with the intervention. Scores range from 8 to 32, with higher scores indicating greater satisfaction with the intervention.
Insomnia Severity Index (ISI) | Post intervention (final study visit)
  The Insomnia Severity Index (ISI) is a seven-item questionnaire developed to assess the severity of insomnia symptoms. Scores range from 0 to 28, with higher scores indicating more severe symptoms.
Pittsburgh Sleep Quality Index (PSQI) | Post intervention (final study visit)
  The Pittsburgh Sleep Quality Index (PSQI) is a sleep questionnaire that evaluates seven primary components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction over a one-month period. The PSQI is used to assess the impact of cognitive behavioral therapy for insomnia (CBT-I) on these sleep components. Scores range from 0 to 21, with higher scores indicating poorer sleep quality.
Epworth Sleepiness Scale (ESS) | Post intervention (final study visit)
  The Epworth Sleepiness Scale (ESS) is a sleep questionnaire consisting of 8 items that assesses daytime sleepiness. A score of 10 or higher indicates pathological daytime sleepiness. The total score ranges from 0 to 24, with higher scores indicating greater daytime sleepiness.
Canadian Occupation Performance Measure (COPM) | Post intervention (final study visit)
  The Canadian Occupation Performance Measure (COPM) is a self-reported measure of an individual's perceived performance and satisfaction in important daily activities. Scores range from 1 (low) to 10 (high) for both performance and satisfaction, with higher scores indicating better outcomes.
Activity Card Sort (ACS) | Post intervention (final study visit)
  Occupational therapists use the Activity Card Sort (ACS) to help clients describe their social, instrumental, and leisure activities. For this study, we are going to use Electronic Activity Card Sort. It serves the same purpose as the paper/card version but is administered electronically. Total scores are expressed as a percentage (0-100%), with higher scores indicating greater participation and activity engagement.

SECONDARY OUTCOMES:
Dysexecutive Questionnaire (DEX) | Baseline (day 1)
  The Dysexecutive Questionnaire (DEX) is a self- or informant-reported measure of everyday executive function difficulties, including problems with planning, organization, problem-solving, and behavior regulation. Total scores range from 0 to 80, with higher scores indicating more pronounced executive dysfunction.
Neurobehavioral Symptom Inventory (NSI) | Baseline (day 1)
  The Neurobehavioral Symptom Inventory (NSI) is a self-reported measure of common mild Traumatic Brain Injury (mTBI) symptoms, including cognitive, affective, sleep, and somatic complaints. Total scores typically range from 0 to 100, with higher scores reflecting greater symptom severity.
Fatigue Severity Scale (FSS) | Baseline (day 1)
  The Fatigue Severity Scale (FSS) is a self-administered instrument designed to evaluate the impact of fatigue on daily functioning. It consists of 9 items, each rated on a scale from 1 to 7, yielding a total score of 9 to 63. Higher average scores reflect greater fatigue severity.
Beck's Depression Inventory (BDI) | Baseline (day 1)
  The Beck Depression Inventory-II (BDI-II) is a self-reported questionnaire assessing the severity of depressive symptoms over the past two weeks. Total scores range from 0 to 63, with higher scores reflecting more severe depression.
Depression Anxiety Stress Scale (DASS) | Baseline (day 1)
  The Depression Anxiety Stress Scale- 21 Items (DASS-21) is a self-reported questionnaire measuring symptoms of depression, anxiety, and stress over the past week. Each subscale (Depression, Anxiety, Stress) is scored from 0 to 63, with higher scores reflecting more severe symptoms.
Quality of Life after Brain Injury (QOLIBRI) | Baseline (day 1)
  The Quality of Life after Brain Injury (QOLIBRI) is a self-reported measure assessing health-related quality of life in individuals after traumatic brain injury, across physical, cognitive, emotional, and social domains. Total scores range from 0 to 100, with higher scores reflecting better quality of life.
Dysexecutive Questionnaire (DEX) | Post intervention (final study visit)
  The Dysexecutive Questionnaire (DEX) is a self- or informant-reported measure of everyday executive function difficulties, including problems with planning, organization, problem-solving, and behavior regulation. Total scores range from 0 to 80, with higher scores indicating more pronounced executive dysfunction.
Neurobehavioral Symptom Inventory (NSI) | Post intervention (final study visit)
  The Neurobehavioral Symptom Inventory (NSI) is a self-reported measure of common mild Traumatic Brain Injury (mTBI) symptoms, including cognitive, affective, sleep, and somatic complaints. Total scores typically range from 0 to 100, with higher scores reflecting greater symptom severity.
Fatigue Severity Scale (FSS) | Post intervention (final study visit)
  The Fatigue Severity Scale (FSS) is a self-administered instrument designed to evaluate the impact of fatigue on daily functioning. It consists of 9 items, each rated on a scale from 1 to 7, yielding a total score of 9 to 63. Higher average scores reflect greater fatigue severity.
Beck's Depression Inventory (BDI) | Post intervention (final study visit)
  The Beck Depression Inventory-II (BDI-II) is a self-reported questionnaire assessing the severity of depressive symptoms over the past two weeks. Total scores range from 0 to 63, with higher scores reflecting more severe depression.
Depression Anxiety Stress Scale (DASS) | Post intervention (final study visit)
  The Depression Anxiety Stress Scale- 21 Items (DASS-21) is a self-reported questionnaire measuring symptoms of depression, anxiety, and stress over the past week. Each subscale (Depression, Anxiety, Stress) is scored from 0 to 63, with higher scores reflecting more severe symptoms.
Quality of Life after Brain Injury (QOLIBRI) | Post intervention (final study visit)
  The Quality of Life after Brain Injury (QOLIBRI) is a self-reported measure assessing health-related quality of life in individuals after traumatic brain injury, across physical, cognitive, emotional, and social domains. Total scores range from 0 to 100, with higher scores reflecting better quality of life.

OTHER OUTCOMES:
Montreal Cognitive Assessment (MoCA) | The instrument will be used to assess the study's eligibility and inclusion/exclusion criteria prior to study initiation.
  The Montreal Cognitive Assessment (MoCA) is a brief cognitive screening tool that assesses multiple cognitive domains including memory, attention, language, visuospatial skills, and executive function. Total scores range from 0 to 30, with higher scores reflecting better overall cognitive performance.
Patient Health Questionnaire-9 (PHQ-9) | The instrument will be used to assess the study's eligibility and inclusion/exclusion criteria prior to study initiation.
  The Patient Health Questionnaire-9 (PHQ-9) is a self-reported measure assessing the severity of depressive symptoms over the past two weeks. Total scores range from 0 to 27, with higher scores reflecting more severe depression.
Generalized Anxiety Disorder-7 (GAD-7) | The instrument will be used to assess the study's eligibility and inclusion/exclusion criteria prior to study initiation.
  The Generalized Anxiety Disorder-7 (GAD-7) is a self-reported questionnaire assessing the severity of generalized anxiety symptoms over the past two weeks. Total scores range from 0 to 21, with higher scores reflecting more severe anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boone AE, Henderson WL, Zenoozi S. Surveying the Landscape of Persistent Concussive Symptoms in Adults Through an Occupational Lens. Am J Occup Ther. 2024 Mar 1;78(2):7802180190. doi: 10.5014/ajot.2024.050405. PMID 38373065